CLINICAL TRIAL: NCT05876611
Title: Clinical Application of a Self Stabilizing Atlantoaxial Fusion Cage: a Cohort Study
Brief Title: Clinical Application of a Self Stabilizing Atlantoaxial Fusion Cage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZL 2022 1 0362717.5
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-05

CONDITIONS: Atlantoaxial Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Using the new type of self stabilizing atlantoaxial fusion cage: Use the new type of self stabilizing atlantoaxial fusion cage to treat atlantoaxial dislocation.
  Interventions: Device: New type of self stabilizing atlantoaxial fusion cage
- Using other fusion systems: Use screw and plate system or other existing models of fusion cages.

INTERVENTIONS:
Device: New type of self stabilizing atlantoaxial fusion cage — Using the above-mentioned new fusion cage for the treatment of atlantoaxial dislocation
  Groups: Using the new type of self stabilizing atlantoaxial fusion cage

SUMMARY:
Conventional open surgery often requires extensive dissection of the muscle insertion points of the suboccipital muscle group during the insertion position and direction of the atlas axis screw, resulting in sustained postoperative occipital neck pain and movement dysfunction. In order to overcome the shortcomings of the prior art mentioned above, the present invention provides a self stabilizing fusion cage with a wing plate. During surgery, a thinner and smaller screw through the wing plate is used to achieve a secure connection between the atlas axis and the fusion cage. Due to the smaller screw size, the screw placement has higher safety. The purpose of this study is to compare the advantages of using this new fusion cage compared to traditional surgical instruments.

ELIGIBILITY:
Inclusion Criteria:

1. Atlantoaxial dislocation
2. Agree to use a new self stabilizing atlantoaxial fusion cage for surgery where feasible
3. Sign an informed consent form;

Exclusion Criteria:

1. Atlantoaxial dislocation without surgical treatment
2. Patients who refuse to participate in this project

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with atlantoaxial dislocation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
fusion rate | 12 month follow up
  Postoperative atlantoaxial fusion conditions
neural functions | 12 month follow up
  Postoperative neurological function recovery conditions
complications | 12 month follow up
  Short or long-term postoperative complications